CLINICAL TRIAL: NCT03297008
Title: Understanding Innate and Adaptive Immunological Response in Stool and Saliva Samples in Healthy Donors
Brief Title: Biomarkers in Saliva and Stool
Status: Terminated | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO-MK-001
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: healthy; saliva; stool; biomarkers; Respiratory Syncytial Virus; Rotavirus; Immunoglobulin; Antibody

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva, Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No internvetion — No intervention, this is an observational study

SUMMARY:
To collect saliva and stool samples using the salimetrics swab and self-stool collection kit, process and store samples in a standardized manner. Following this, perform immunological assays such as enzyme-linked immunosorbent assay, multiplex bead assay and Immunocap to correlate the salivary and fecal levels of biomarkers in healthy donors. As this method is non-invasive, we believe that more people will be willing to donate samples.

DETAILED DESCRIPTION:
Many soluble factors found in blood can be detected in saliva and stool. Often levels of these factors are found to correlate between body fluids, though the exact relationship between systemic (blood) and local (saliva and stool) immunity is not well established yet. Saliva- and stool-associated factors are produced in the oral cavity and in the gut, which represent mucosal sites that potentially come in direct contact with pathogens. Thus, the levels of mucosal-associated soluble factors can better represent the local immune response at these sites.

It is becoming clear now that saliva and stool can be used to analyze inflammatory responses as well. In a recent study, 20 possible salivary biomarkers related to obesity were surveyed and the authors found four biomarkers that exhibit significant change with increasing body weight in a pediatric population. Salivary C-reactive protein (CRP), salivary insulin, leptin and adiponectin were found to be different in obese children compared to healthy normal weight children. This data suggests that saliva could be a useful blood surrogate for the study of metabolic complications of obesity in children, where repeated blood sampling can be both traumatic and difficult. The results of this study also provide insight into the early development of metabolic disease in children. (Goodson, Kantarci et al. 2014). In another study, cytokines-chemokines-growth factors (CCGFs) were measured using multiplex bead assays and compared between plasma, saliva and urine collected from 20 male and female healthy volunteers. By analyzing more than one sample types from the same subject would increase the possibility of identifying biomarker(s) for any inflammatory disease. In this study, gender-specific CCGFs were also observed and concentrations of some CCGFs varied between genders. This information is also valuable for biomarker discovery that by combining male and female subjects in a clinical trial would eliminate false discovery of biomarkers (Khan 2012).

The mucosal immune system can be also understood by analyzing stool samples. In a recent study, it is shown that a particular bacterial predominance, such as Bifidobacterium sp., may enhance thymic development and immune responses to both oral and parenteral vaccines early in infancy, whereas a deviation from this pattern, resulting in greater bacterial diversity, may cause systemic inflammation (neutrophilia) and lower vaccine responses. Thus, vaccine responsiveness may be improved by promoting intestinal Bifidobacteria sp. and minimizing dysbiosis early in infancy (Huda, Lewis et al. 2014). Of note, the hallmark of adequate mucosal immune responses is the production of secretory immunoglobulin A (SIgA), which can prevent infection and remove antigen crossing the mucosal barrier.SIgAis also imperative to establish mutualism between host and the intestinal microbiota (Maynard, Elson et al. 2012). Hence measurement of SIgA can help to assess the mucosal immunity.

Despite saliva and stool samples are increasingly studied in order to assess mucosal immune response and/or clinical outcomes, there is still a lack of established methodology to be routinely used in diagnostic laboratories and clinical trials. Therefore our aim is to collect saliva and stool samples using the salimetrics swab and self-stool collection kit from a cohort of 60 volunteers, process and store samples in a standardized manner. Following this, we intend to perform immunological assays such as enzyme-linked immunosorbent assay, multiplex bead assay and Immunocap to correlate the salivary and fecal levels of biomarkers in healthy donors. As this method is non-invasive, we believe that more people will be willing to donate samples. It is also easy to self-collect and it is cost efficient.

ELIGIBILITY:
Inclusion Criteria:

• Healthy volunteers of age 0-60 years old

Exclusion Criteria:

* Volunteers with any known infectious diseases, such as HIV and Hepatitis B
* Volunteers with any acute or chronic illness, such as chronic inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis)
* Volunteers with oral diseases/ulcers

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Volunteers in Singapore between 0 and 60 years of age
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Establish methods to detect immune markers in non-invasive samples: Saliva and stool in healthy volunteers | 1 year after completion of recruitment
  ELISA RSV specific Immunoglobulin in saliva
Establish methods to detect immune markers in non-invasive samples: Saliva and stool in healthy volunteers | 1 year after completion of recruitment
  ELISA Rotavirus specific Immunoglobulin in stool

SECONDARY OUTCOMES:
Difference in RSV-specific Immunoglobulins between age groups. | 1 year after completion of primary outcome
  Correlation between age and RSV-specific Immunoglobulins in saliva
Difference in RSV-specific Immunoglobulins between age groups. | 1 year after completion of primary outcome
  Correlation between age and rotavirus-specific Immunoglobulins in stool

OTHER OUTCOMES:
Establish methods to detect immune markers in non-invasive samples: Saliva and stool in healthy volunteers | 1 year after completion of primary outcome
  ELISA RSV specific Immunoglobulin in stool
Establish methods to detect immune markers in non-invasive samples: Saliva and stool in healthy volunteers | 1 year after completion of primary outcome
  ELISA Rotavirus specific Immunoglobulin in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sandalova, PhD, Principal Investigator — Nutricia Research
Locations (1):
- Danone Nutricia Research, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
IDP is not going to be shared.